CLINICAL TRIAL: NCT03575481
Title: Differences in Muscle Activity and Fatigue of the Upper Limb Between Task-Specific Training and Robot Assisted Training Among Individuals Post Stroke
Brief Title: Muscle Activity of the Upper Limb Between Task-Specific and Robot Assisted Training Among Individuals Post Stroke
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Sponsor
Other Study IDs: 0295-15-HMO
Record Dates: First submitted 2018-06-17; First posted 2018-07-02 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post stroke patients
  Interventions: Diagnostic Test: The RAT and The TST

INTERVENTIONS:
Diagnostic Test: The RAT and The TST — The RAT (ReoGo; Motorika Medical, Caesarea, Israel) The TST protocol included the conventional, repetitive, task-oriented training of the affected arm.

SUMMARY:
The investigators compared the activity and fatigue of upper extremity muscles, pain levels, subject satisfaction levels, perceived exertion, and number of repetitions in Task-Specific Training (TST) compared with Robot-Assisted Training (RAT) in individuals post-stroke.

DETAILED DESCRIPTION:
Twenty sub-acute post stroke subjects received one TST and one RAT. They marked the pain level in their paretic extremity before and after each session. Muscle activity levels and fatigue and number of repetitions were monitored during each session. The subjective assessment questionnaire of treatment and the Borg scale were administered post-session.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 85 year old individuals up to three months following stroke
* National Institutes of Health Stroke Scale (NIHSS) score 3-15
* Intact cognitive function
* mild to moderate weakness of the affected hand
* normal or corrected eyesight

Exclusion Criteria:

* neurological, cardio-vascular or orthopedic impairment, unrelated to the stroke, which restricts upper limb function
* a pace-maker

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stroke survivors
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
Muscle activity | 30 minutes
  The activity levels of electromyographic signal (in millivolts) will be averaged for the duration of the recording.
Muscle fatigue | 30 minutes
  Fatigue expressed by calculation of the the difference between the median frequency in the first 5 minutes and last five minutes of a 30 minute session

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No